CLINICAL TRIAL: NCT04336683
Title: Feasibility Study for Ultrasound-Guided Interstitial Brachytherapy for Gynecological CancersV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 106088
Record Dates: First submitted 2020-03-10; First posted 2020-04-07 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Gynecologic Cancer
Keywords: 3D Ultrasound; Intervention
MeSH Terms: interventions — Brachytherapy

STUDY DESIGN:
Intervention Model Description: Patients who are assigned to gynecological brachytherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Other): Patients undergoing gynecological brachytherapy, will be imaged with a 3D ultrasound medical device for the purpose of efficacy testing.
  Interventions: Device: Interstitial and intracavitary brachytherapy

INTERVENTIONS:
Device: Interstitial and intracavitary brachytherapy — Standard of care in interstitial or intracavitary brachytherapy is to insert the brachytherapy needle and applicator with no standard real-time image guidance. Interstitial brachytherapy is done under general anesthesia. Trans-abdominal and trans-rectal standard 2D ultrasound is used in some cases, but is typically not consistent and therefore its value is limited. Pre-procedure imaging in the form of MRI is used to help guide needles insertion as well as the clinical exam. Post-procedure CT is done for radiation planning

SUMMARY:
Brachytherapy treatment in gynecological cancers is an essential component to delivering adequate doses of radiation to a tumour while sparing normal tissue. Interstitial and intracavitary brachytherapy is often needed in advanced or recurrent disease, in cases where intrauterine brachytherapy may not deliver the optimal outcome. Interstitial brachytherapy is based on a defined template-and-needle system, and the procedure relies on clinical examination and pre-treatment imaging to guide needle insertion. There is currently no standard image-guided process to help direct needles in the pelvis. The investigators propose a 3D ultrasound device that will provide real-time imaging for the brachytherapy procedure which will aid in avoiding needle insertion into pelvic organs and result in optimal dose coverage to the tumour.

DETAILED DESCRIPTION:
This is an efficacy study to optimize the use of three-dimensional ultrasound imaging for interstitial and intracavitary brachytherapy. In this study, 3DUS images will be acquired during the regular clinical procedure to assess the quality of the images, anatomical detail and location of needles. The acquired images will be analyzed post-treatment and fused with pre-treatment MRI, and post-treatment CT scans to develop a virtual simulated radiation treatment plan, and to verify the applicator positions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or recurrent gynecological malignancies who are offered interstitial or intracavitary brachytherapy treatment. These typically would include patients with primary or recurrent vaginal cancers, endometrial cancers or cervical cancers. Histologies of these cancers are typically adenocarcinomas or squamous cell carcinomas

Exclusion Criteria:

* Above patients who are not offered interstitial or intracavitary brachytherapy as a treatment modality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females patients with locally advanced or recurrent gynecological malignancies who are offered interstitial or intracavitary brachytherapy treatment.
Enrollment: 35 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of the 3DUS device to visualize applicators | 16 Weeks
  The number of applicators identified within the 3D ultrasound image.

SECONDARY OUTCOMES:
3DUS to CT Fusion | 16 Weeks
  DICE coefficient of the tumour and needle applicators

CONTACTS AND LOCATIONS:
Overall Officials: David D'Souza, MD, Principal Investigator — Schulich School of Medicine and Dentistry
Locations (1):
- London Regional Cancer Program, Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodgers JR, Hrinivich WT, Surry K, Velker V, D'Souza D, Fenster A. A semiautomatic segmentation method for interstitial needles in intraoperative 3D transvaginal ultrasound images for high-dose-rate gynecologic brachytherapy of vaginal tumors. Brachytherapy. 2020 Sep-Oct;19(5):659-668. doi: 10.1016/j.brachy.2020.05.006. Epub 2020 Jul 3. PMID 32631651
- [Result] Rodgers JR, Bax J, Surry K, Velker V, Leung E, D'Souza D, Fenster A. Intraoperative 360-deg three-dimensional transvaginal ultrasound during needle insertions for high-dose-rate transperineal interstitial gynecologic brachytherapy of vaginal tumors. J Med Imaging (Bellingham). 2019 Apr;6(2):025001. doi: 10.1117/1.JMI.6.2.025001. Epub 2019 Apr 8. PMID 30989088
- [Result] Rodgers JR, Mendez LC, Hoover DA, Bax J, D'Souza D, Fenster A. Feasibility of fusing three-dimensional transabdominal and transrectal ultrasound images for comprehensive intraoperative visualization of gynecologic brachytherapy applicators. Med Phys. 2021 Oct;48(10):5611-5623. doi: 10.1002/mp.15175. Epub 2021 Sep 2. PMID 34415069